CLINICAL TRIAL: NCT03849027
Title: MethOxyflUraNe at moderaTe High AltItudes for PAIN Management: A Randomised, Double-blind, Cross-over Study
Brief Title: MethOxyflUraNe at moderaTe High AltItudes for PAIN Management
Acronym: MOUNTAIN-PAIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Ross Hofmeyr, Prof, University of Cape Town
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MOUNTAIN-PAIN
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Pain
Keywords: altitude; analgesia; methoxyflurane; wilderness medicine
MeSH Terms: conditions — Pain; Agnosia | interventions — Methoxyflurane

STUDY DESIGN:
Intervention Model Description: randomised, controlled, cross-over
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methoxyflurane (Experimental): Inhaled methoxyflurane once-off dose of 3 ml will be administered via the inhaler at each dosing visit .
  Inhaled methoxyflurane will be administered using the disposable field inhaler device (Penthrop®).
  Interventions: Drug: Methoxyflurane
- Sham Methoxyflurane (Sham Comparator): The sham inhaler will have one droplet of methoxyflurane applied to the outer surface, but no drug in the vaporization chamber to give off the prominent odour with no analgesic effect, partially blinding the participants to the test
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methoxyflurane — Inhaled methoxyflurane will be administered using the disposable field inhaler device (Penthrop®) according to the recommended dosing schedule.
  Other Names: Penthrop; Penthrox
  Arms: Methoxyflurane
Drug: Placebo — The sham inhaler will have one droplet of methoxyflurane applied to the outer surface, but no drug in the vaporization chamber to give off the prominent odour with no analgesic effect, partially blinding the participants to the test.
  Other Names: Sham methoxyflurane
  Arms: Sham Methoxyflurane

SUMMARY:
A randomised, double-blind, cross-over study to assess the analgesic effect of methoxyflurane at moderate high altitudes in a wilderness field setting.

Phase IV, randomised, double-blind, cross-over clinical trial to evaluate the analgesic effect of methoxyflurane at moderate high altitudes in a wilderness field setting, in 24 healthy volunteers

DETAILED DESCRIPTION:
Primary outcome: To assess the analgesic efficacy of inhaled methoxyflurane at moderate high altitudes in a wilderness setting.

Secondary outcomes: To assess the comparative safety and adverse events with inhaled methoxyflurane at moderate high altitudes in a wilderness setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 65 years of age (inclusive).
2. Able to provide informed consent and comply with study-related procedures

Exclusion Criteria:

1. History of diabetes
2. Renal or hepatic disease or impairment (defined as a value exceeding the maximum reference range)
3. Chronic or nociplastic pain
4. Chronic fatigue syndrome
5. Chronic/regular use of analgesic medications
6. Personal or familial history of malignant hyperthermia
7. Personal or familial history of anaesthesia-induced rhabdomyolysis
8. Personal history of anaesthesia volatile-induced hepatitis or drug induced liver injury
9. Recent volatile anaesthesia (within 6 months)
10. History of significant altitude-related illness
11. Significant underlying medical condition which precludes gentle exercise at moderate high altitude (<2500 m ASL) as determined by the investigators
12. Hypersensitivity to Penthrox/Penthrop®, methoxyflurane or any fluorinated anaesthetic.
13. Concurrent treatment with CYP 2A6 or CYP 2E1 enzyme inducers (such as: phenobarbital, rifampicin, alcohol or isoniazid)
14. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Analgesic effect | Up to 3 weeks
  Percentage change in analgesic effect between methoxyflurane inhalation at sea level (ALT 0) and 2250m (ALT 2; moderate high altitude).

SECONDARY OUTCOMES:
Safety and adverse events | Up to 3 weeks
  Comparative safety and adverse events with inhaled methoxyflurane at moderate high altitudes in a wilderness setting

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hofmeyr, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town Department of Anaesthesia & Perioperative Medicine, Cape Town, Western Cape, South Africa